CLINICAL TRIAL: NCT06625840
Title: A Randomized, Double-Blind Clinical Trial to Assess the Safety, Tolerability, and Pharmacokinetics of MK-1167 in Healthy Elderly Participants
Brief Title: A Study of MK-1167 in Healthy Elderly Participants (MK-1167-004)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1167-004; MK-1167-004 (Other: MSD)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Panel A (Experimental): Participants receive a loading dose of MK-1167 or Placebo orally on day 1, followed by a once daily (QD) maintenance dose orally on days 2 to 16.
  Interventions: Drug: MK-1167; Drug: Placebo
- Panel B (Experimental): Participants receive a loading dose of MK-1167 or Placebo orally on days 1 to 3, followed by a QD maintenance dose orally on days 4 to 16.
  Interventions: Drug: MK-1167; Drug: Placebo

INTERVENTIONS:
Drug: MK-1167 — Oral Administration
Drug: Placebo — Oral Administration

SUMMARY:
The goal of this study is to learn how safe MK-1167 is in healthy elderly adults and how well people tolerate it.

ELIGIBILITY:
The main inclusion criteria include but are not limited to the following:

* Be in good health

The main exclusion criteria include but are not limited to the following:

* History of clinically significant endocrine, GI, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases.
* History of cancer (malignancy).

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing an Adverse Event (AE) | Up to approximately 41 days
  An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study treatment. For each arm, the number of participants experiencing an AE will be assessed.
Number of Participants Discontinuing Study Treatment due to an AE | Up to approximately 16 days
  An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study treatment. For each arm, the number of participants experiencing an AE will be assessed.
Area Under the Concentration-Time Curve from 0 to 24 hours (AUC0-24) of MK-1167 after Multiple Doses | Predose and at designated timepoints up to 24 hours postdose on days 1, 8 and 16
  Blood samples will be collected to determine the AUC0-24 of MK-1167.
Maximum Concentration (Cmax) of MK-1167 after Multiple Doses | Predose and at designated timepoints up to 24 hours postdose on days 1 and 8 and up to 600 hours postdose on day 16
  Blood samples will be collected to determine the Cmax of MK-1167.
Concentration at 24 hours (C24) of MK-1167 after Multiple Doses | 24 hours postdose on days 1, 8 and 16
  Blood samples will be collected to determine the C24 of MK-1167.
Time to reach maximum concentration (Tmax) of MK-1167 after Multiple Doses | Predose and at designated timepoints up to 24 hours postdose on days 1 and 8 and up to 600 hours postdose on day 16
  Blood samples will be collected to determine the Tmax of MK-1167.
Apparent Clearance (CL/F) of MK-1167 after Multiple Doses | Predose and at designated timepoints up to 600 hours postdose on day 16
  Blood samples will be collected to determine the CL/F of MK-1167.
Volume of Distribution (Vz/F) of MK-1167 at Steady State after Multiple Doses | Predose and at designated timepoints up to 600 hours postdose on day 16
  Blood samples will be collected to determine the Vz/F of MK-1167.
Apparent Half Life (t½) of MK-1167 after Multiple Doses | Predose and at designated timepoints up to 600 hours postdose on day 16
  Blood samples will be collected to determine the t½ of MK-1167.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- California Clinical Trials Medical Group managed by PAREXEL-PAREXEL International (Site 0001), Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com